CLINICAL TRIAL: NCT01092806
Title: Effects on Insulin Secretion and Sensitivity of Two Different Formulations Tacrolimus - Prograf® and Advagraf®
Brief Title: Insulin Secretion and Advagraf
Acronym: ADVA-09
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anders Åsberg, Study leader, University of Oslo School of Pharmacy
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ADVA-09
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Post Transplant Diabetes Mellitus
Keywords: tacrolimus; pharmacokinetics; formulations; once daily; twice daily; renal transplant recipients; Kidney transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prograf (Active Comparator): Patients are treated until steady-state conditions with Prograf and then investigated with clamp
  Interventions: Drug: Tacrolimus
- Advagraf (Experimental): The patients are treated with Advagraf until steady-state conditions and then investigated with clamp
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Two different formulations of the drug is compared. The dose is adjusted according to whole blood concentrations in accordance with center protocol. Switch between the two formulations are done by a 1:1 conversion of daily dose.
  Other Names: Prograf (BID formulation); Advagraf (QD formulation)

SUMMARY:
One of the main side-effects of tacrolimus in solid organ transplanted patients is post transplant diabetes mellitus (PTDM). It is not known if different pharmacokinetic properties influence the risk of developing PTDM. It is possible that it either is high peak concentrations of high overall systemic exponation that is responsible for the effect on insulin secretion. With the new slow-release formulation of tacrolimus (Advagraf) a different pharmacokinetic profile is introduced to patients and it is of interest to investigate if this affects insulin secretion and insulin sensitivity of patients.

Hypothesis: The pharmacokinetic profile of tacrolimus affects the insulin secretion in renal transplant recipients.

DETAILED DESCRIPTION:
Study objectives

The primary objective is to compare insulin secretion (Secr2.phase) between the two different formulations of Tac.

Secondary objectives are to compare the effect of the two formulations on Secr1.phase, insulin sensitivity and to investigate possible associations with individual systemic tacrolimus exposures.

Study design

Twenty adult kidney transplanted patients treated with Prograf® twice daily or Advagraf® once daily will be included in the study. Eligible patients may be included in a stable posttransplant phase (no Tac dose adjustments or acute rejection episodes the preceding 2 weeks). A 3-hour hyperglycaemic clamp will be performed while patients are treated with their standard Tac formulation and repeated 4-6 weeks after switching to the alternative Tac formulation. The clamp investigation will be done after administration of the morning dose of Tac. Samples for measurement of Tac whole blood concentrations will be drawn for all patients up to 24 hours after morning Tac dosing. It is not mandatory for all patients to perform full 24 hour pharmacokinetic investigations.

Switching to the alternative Tac formulation will be performed in a 1:1 daily dose ratio and subsequently adjusted according to centre protocol for trough concentrations (5-10 ng/mL). Patients will meet for trough concentration measurements at Rikshospitalet for appropriate dose adjustment in the period between the two investigations days.

Patients

The patients will primarily be recruited from the great-Oslo area and all study visits will be performed at Rikshospitalet. Patients will otherwise follow standard post transplant procedures at their local hospital during the study period. Patients included in other clinical trials are also eligible for inclusion in the present study as long as they are not treated with investigational drugs.

Informed consent will be obtained according to the Declaration of Helsinki and ICH-GCP guidelines. Patients and investigator will sign the patient information which will be kept on file. The patient will receive a copy of the patient information. Patient data will be recorded in Case Report Forms (CRF) and all information will be handled confidentially. Any complications will be recorded.

Glucose clamp calculations

Lean body mass (lbm) is estimated using Hume's formula [12] which correlates well with tritiated water or electrical bioimpedance measures [13]. Secr1.phase is calculated as the area under serum insulin vs. time curve (AUC, trapezoidal rule) during the first 10 min of the clamp procedure, and Secr2.phase is calculated as the insulin AUC during the last hour (120-180 min) of the clamp procedure. The same calculations were also performed for C-peptide concentrations. Glucose disposal rate (GDR) is calculated from the amount of glucose infused during the last hour of the clamp. The IS index (ISI) is calculated as GDR [mmol/kg (lbm)*min] divided by mean serum insulin (pmol/l) in the same period. Glucose clearance is calculated as ISI divided by mean serum glucose during the last 60 min of the clamp [14].

Pharmacokinetic calculations

Nonlinear mixed effects modeling (NONMEM software version VI and Intel Fortran (version 8) compilation tool) will be used to analyze the dose-concentration-time data for Tac using a population approach. The pharmacokinetic profile data will be used to develop a pharmacokinetics model including the effect of major covariates (e.g. age, gender, body size, renal function, hematocrit, acute rejection status etc.) on CL/F and V/F from the 24-hour pharmacokinetics investigations. If applicable additional trough concentration data from the routine follow-up of the patients in the study will be used to develop the model.

Exclusion of patient data will only be allowed if Tac concentrations have not been able to be measured accurately or in case of unavailable information that may interfere with pharmacokinetic evaluation, e.g. exact blood sampling time or dose given.

The POSTHOC, MAXEVAL=0 option in NONMEM will be used to estimate individual AUC0-24 and half-lives for each individual. Actually measured Ctrough, Cmax and Tmax values will also be used to describe the pharmacokinetic properties of the patients.

Statistical considerations

Sample size:

Based on the assumption that a 15% relative change in insulin secretion between the two formulations are clinically relevant and a relative standard deviation of 25% 20 patients are needed to assure a power of 80% at a 5% significance level. Patients that drop-out during the study will be substituted.

Analysis plan:

The primary end-point will be analyzed per-protocol by comparing the ratio of insulin sensitivity (Secr2.phase) for the two formulations. Data will be transformed to obtain normal distribution if appropriate.

Secondary endpoints will be analyzed as follows:

* Insulin Secr1.phase
* Insulin sensitivity index (ISI)
* Association between insulin Secr2.phase, Secr1.phase and ISI and systemic exposure of Tac (derived from individual NONMEM estimations)
* All analysis above also performed for C-peptide

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients on stable Tac based immunosuppressive therapy.
* 18 years of age or older.
* Stable prednisolone dose of 5 mg/day or less.
* S-creatinine below 150 umol/L.
* Signed informed consent.

Exclusion Criteria:

* Acute rejection episodes within the last 2 weeks prior to inclusion.
* Changes in Tac dosing within the last 2 weeks prior to inclusion.
* Diabetes mellitus (WHO criteria).
* Pregnant or nursing mothers or women of childbearing potential without acceptable contraception strategy.
* Concomitant treatment with: diltiazem, verapamil, fenytoin, carbamazepine, fluconazole, ketoconazole, voriconazole, erythromycin, clarithromycin.
* Patients treated with investigational drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The primary objective is to compare insulin secretion (Secr2.phase) between the two different formulations of Tac. | 1 month
  Insulin secretion is investigated by hyperglycemic clamp

SECONDARY OUTCOMES:
Secondary objectives are to compare the effect of the two formulations on Secr1.phase, | 1 month
  First phase insulin secretion is investigated by hyperglycemic clamp
insulin sensitivity | 1 month
  Investigated by hyperglycemic clamp

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Midtvedt, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo univeristy hospital, Rikshospitalet, Oslo, Norway